CLINICAL TRIAL: NCT01488448
Title: A Double-Blind, Controlled, Randomized Clinical Trial of Nebulized Hypertonic Saline for Hospitalized Infants With Viral Bronchiolitis
Brief Title: A Study of Hypertonic Saline for Infants Hospitalized With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Alyssa Silver, Attending Physician, Pediatric Hospitalist, Assistant Professor of Pediatrics, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-09-329
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Bronchiolitis
Keywords: Hypertonic saline; Bronchiolitis; Infants; Wheezing; Nebulized; Bronchodilator
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds | interventions — Sodium Chloride; Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebulized Hypertonic Saline (Experimental): 4mL nebulized 3% sodium chloride every 4 hours until discharge
  Interventions: Drug: 3% sodium chloride
- Nebulized Normal Saline (Placebo Comparator): 4 mL nebulized 0.9% sodium chloride every 4 hours until discharge
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: 3% sodium chloride — 4 milliliters delivered via nebulizer with 5 Liters O2 flow every 4 hours until discharge
  Other Names: hypertonic saline; HS
  Arms: Nebulized Hypertonic Saline
Drug: 0.9% sodium chloride — 4 milliliters delivered via nebulizer with 5 Liters O2 flow every 4 hours until discharge
  Other Names: normal saline; NS
  Arms: Nebulized Normal Saline

SUMMARY:
The purpose of this study is to determine if nebulized hypertonic saline (or extra salty water mist) helps infants less than 12 months old hospitalized with bronchiolitis (or bad chest colds) get better enough to be discharged from the hospital sooner than those infants given nebulized normal saline (or regular salty water mist).

DETAILED DESCRIPTION:
Bronchiolitis is a common admitting diagnosis for children less than 1 year of age. Although bronchiolitis has a high prevalence, there is a lack of a unified inpatient treatment plan beyond supportive care of supplemental oxygen and intravenous hydration. There have been many different approaches to the treatment of bronchiolitis, but none have conclusively proven to be beneficial. Several early studies show promise for the use of nebulized hypertonic saline, however the majority of these studies are done outside the United States and with adjunctive therapy. To date, the data suggesting that nebulized hypertonic saline is safe and effective for reducing length of stay in bronchiolitis is strong but not generalizable for the United States. The objective of this study is to conduct the first double-blind, randomized controlled trial in the United States of nebulized hypertonic saline without adjunctive therapy, including infants with bronchiolitis, including those with prior history of wheeze, to assess the effect on length of stay and therefore resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-12 months of age admitted to the hospital with a diagnosis of bronchiolitis.

Exclusion Criteria:

* status asthmaticus
* chronic cardiopulmonary disease
* Trisomy 21
* immunodeficiency or transplant recipient
* neuromuscular disease
* admission directly to the intensive care unit
* previous use of nebulized hypertonic saline less than 12 hours prior to presentation
* previous enrollment in the study in the 72 hours prior to presentation

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa H Silver, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

REFERENCES:
- [Derived] Silver AH, Esteban-Cruciani N, Azzarone G, Douglas LC, Lee DS, Liewehr S, Nazif JM, Agalliu I, Villegas S, Rhim HJ, Rinke ML, O'Connor K. 3% Hypertonic Saline Versus Normal Saline in Inpatient Bronchiolitis: A Randomized Controlled Trial. Pediatrics. 2015 Dec;136(6):1036-43. doi: 10.1542/peds.2015-1037. Epub 2015 Nov 9. PMID 26553190

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertonic Saline: 4 mL nebulized 3% sodium chloride every 4 hours until discharge
- Normal Saline: 4 mL nebulized 0.9% sodium chloride every 4 hours until discharge
Period: Overall Study
Arm/Group | Hypertonic Saline | Normal Saline
Started | 113 | 114
Completed | 93 | 97
Not Completed | 20 | 17
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 9 | 4
Not completed — Physician Decision | 4 | 9
Not completed — Protocol Violation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | Normal Saline | Total
Number analyzed (Participants) | 113 | 114 | 227
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.86 (3.01) | 4.39 (2.95) | 4.1 (2.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 42 | 78
  Male | 77 | 72 | 149

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in the Study-LOS--Intention to Treat Analysis
Description: Length of stay will be defined by the duration between the time of first study treatment to the time a discharge order is placed. Alternatively, if a patient remains inpatient for other, non-bronchiolitis related reasons (i.e. social reasons, etc.) the time a patient could be discharged from the standpoint of bronchiolitis as documented by the attending, will be used.
Time Frame: Time of first study treatment until time of discharge
Population: Intention to Treat Analysis
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 111 | 111
Days | 2.1 [1.2 to 4.6] | 2.1 [1.2 to 3.8]
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Readmission for Bronchiolitis Within 7 Days of Discharge
Description: Phone call at 7 days to assess for readmission to any hospital
Time Frame: within 7 days of hospital discharge
Population: This population is those who completed the study.
Measure: Number; unit: participants
Arm/Group | Nebulized Hypertonic Saline | Nebulized Normal Saline
Number analyzed (Participants) | 93 | 97
participants | 4 | 3
Statistical Analysis 1: Comparison: Nebulized Hypertonic Saline vs Nebulized Normal Saline; Test type: Superiority or Other; p = 0.77, Fisher Exact

3. Secondary Outcome: Clinical Worsening
Description: transfer to the Pediatric Intensive Care Unit (PICU) (including withdrawn from the study for bronchodilator administration who were then transferred to the PICU), or Respiratory Distress Assessment Instrument (RDAI) increase of 4 or more points within 30 minutes of a study treatment
Time Frame: though hospitalization/time period receiving study treatment, average 2-3 days
Population: all patients enrolled in the study were analyzed for events related to clinical worsening
Measure: Number; unit: participants
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 113 | 114
participants | 10 | 9
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.97, Fisher Exact

4. Secondary Outcome: Total Adverse Events
Description: Clinical worsening events (defined prior) + 7 day readmissions
Time Frame: Time of enrollment in the study through 1 week after hospital discharge
Measure: Number; unit: adverse events
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 93 | 97
adverse events | 14 | 12
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.67, Fisher Exact

5. Post Hoc Outcome: LOS in Subgroup of Patients With Testing Positive for Respiratory Syncitial Virus (RSV+)
Time Frame: through hospitalization/while receiving study medication, average 2-3 days
Population: This is the population in the study whose RSV testing was positive.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 69 | 59
days | 2.2 [1.6 to 3.8] | 2.0 [1.2 to 3.2]
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)

6. Post Hoc Outcome: LOS in Patients With a History of Previous Wheeze
Time Frame: through hospitalization/while receiving study medication, average 2-3 days
Population: Subgroup of the study population who reported a history of wheezing prior to this admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 14 | 21
days | 1.7 [1.1 to 2.6] | 2.0 [1.2 to 3.2]
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

7. Post Hoc Outcome: LOS Subgroup Analysis of Patients With a History of Prematurity
Time Frame: through hospitalization/while receiving study medication, average 2-3 days
Population: Patients who reported a history of prematurity/whose Gestational age was <37 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 11 | 15
days | 2.9 [1.9 to 3.6] | 2.2 [1.2 to 3.2]

8. Post Hoc Outcome: LOS Analysis for Patients Whose Study Entry Respiratory Distress Assessment Instrument (RDAI) Was Greater Than or Equal to 4 or Who Had Hypoxia <92%
Time Frame: through hospitalization/while receiving study medication, average 2-3 days
Population: Subgroup of patients who had a study entry Respiratory Distress Assessment Instrument (RDAI) of greater than or equal to 4 points OR hypoxia <92% on admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 62 | 67
days | 2.1 [1.3 to 4.1] | 2.1 [1.3 to 3.7]

9. Primary Outcome: Length of Stay in the Study-LOS by Per Protocol Analysis
Description: as for outcome 1
Time Frame: Time of first study treatment until time of discharge
Population: Per protocol analysis (only includes participants who completed the study)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 93 | 97
Days | 2.0 [1.3 to 3.3] | 2.0 [1.2 to 3.0]
Statistical Analysis 1: Comparison: Hypertonic Saline vs Normal Saline; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Normal Saline: 4mL nebulized 0.9% sodium chloride every 4 hours until discharge
Arm/Group | Hypertonic Saline | Normal Saline
Serious Adverse Events (participants affected / at risk) | 13/113 | 10/114
Other Adverse Events (participants affected / at risk) | 0/113 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypertonic Saline (N=113) | Normal Saline (N=114)
Transfer to PICU (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Readmission-respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Readmission-non-respiratory (Investigations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes